CLINICAL TRIAL: NCT06959082
Title: A Multi-center, Randomized, Open-label, Parallel-group, Phase 2 Study to Evaluate the Efficacy and Safety of VS-101 in Combination With Chemoradiotherapy (CRT) in Patients With Head and Neck Cancer
Brief Title: Efficacy and Safety Evaluation of VS-101 in Combination With Chemoradiotherapy in Patients With Head and Neck Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VSPharmTech Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VS-101-C3
Record Dates: First submitted 2025-04-16; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer Squamous Cell Carcinoma
MeSH Terms: interventions — Cisplatin; Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2 mg of VS-101 + CRT (Experimental): 2 mg of VS-101 + CRT
  Interventions: Drug: VS-101; Drug: Cisplatin; Radiation: Radiation
- 5 mg of VS-101 + CRT (Experimental): 5 mg of VS-101 + CRT
  Interventions: Drug: VS-101; Drug: Cisplatin; Radiation: Radiation
- Only CRT (Placebo Comparator): Only CRT
  Interventions: Drug: Cisplatin; Radiation: Radiation

INTERVENTIONS:
Drug: VS-101 — VS-101
  Arms: 2 mg of VS-101 + CRT; 5 mg of VS-101 + CRT
Drug: Cisplatin — Cisplatin
Radiation: Radiation — Radiation

SUMMARY:
This will be a multi-center, randomized, open-label, parallel-group study in adult patients with head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged more than 18 years at the time of ICF signing
2. Diagnosed based on position emission tomography (PET), computed tomography (CT), or magnetic resonance imaging (MRI) with pathologically confirmed (histologic or cytological) head and neck squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx
3. Defined by American Joint Committee on Cancer [AJCC] Guidelines 8th Edition:

   * Oral cavity, hypopharynx, or larynx (independent of p16): Stage III, IVa, IVb per TNM guidelines; or
   * Oropharyngeal p16 negative disease: Stage III, IVa, IVb per TNM guidelines; or
   * Oropharyngeal p16 positive disease: T4 (N0-N3), M0; or N3 (T1-T4), M0.
4. Have measurable disease based on RECIST 1.1
5. Subjects with head and neck cancer who have limited to those receiving definitive CRT without surgical excision
6. Subjects prescribed standard intensity-modulated radiation therapy (IMRT) with daily fractions of 2.0 Gy to a cumulative planned dose of 70 Gy
7. Subjects with Eastern Cooperative Oncology Group (ECOG) Performance Statue (PS) of 0 ~ 2
8. Subjects with the status of National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 Grade 1 or lower for acute or chronic adverse reaction at the time of screening
9. Subjects with an expected survival period of at least 20 weeks
10. Subjects who can comply with the requirements of the clinical trial protocol
11. Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

1. Medical History

   1. Patients with a history of prior radiation to the head and neck region or with a known susceptibility to radiation (e.g., genetic condition, connective tissue disease)
   2. Patients with suicidal behavior, major depression, or other psychiatric disorders (bipolar disorder, attention deficit hyperactivity disorder, etc.)
   3. Patients with neuroleptic malignant syndrome, tardive dyskinesia, elderly with dementia, uncontrolled hyperglycemia and diabetes, and patients with venous thromboembolism
   4. Patients with orthostatic hypotension caused by cardiovascular disease (history of myocardial infarction or ischemic heart disease, heart failure or electrocardiogram abnormality), cerebrovascular disease, or conditions prone to hypotension (dehydration, decreased blood volume, and taking antihypertensive medication)
   5. Patients with a history of seizures
   6. Patients with possible cognitive and motor performance impairments (drowsiness and sedation) (However, if the investigator determines that cognitive and motor performance impairments are not likely to be impaired, enrollment is possible.)
   7. Patients with conditions that may increase core body temperature (such as strenuous exercise, exposure to excessive heat, taking anticholinergic drugs, or patients prone to dehydration)
   8. Patients with dysphagia [those who are taking drugs that may be affected (However, if the investigator determines that dysphagia is unlikely to occur, enrollment is possible), those with aspiration pneumonia, those with esophageal dyskinesia]
   9. Patients with a history of clinically significant allergic disease (with the exception of mild allergic rhinitis that does not require treatment) or hypersensitivity to other drugs(aspirin, antibiotics, etc.)
2. Subjects who show abnormalities in the following test results at the time of screening:

   1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 × upper limit of normal (ULN)
   2. Creatine clearance ≤60 mL/min (using Cockcroft-Gault (C-G) formula)
   3. Absolute neutrophil count (ANC) <1,500/µL
   4. Platelets <100,000/µL
   5. Hemoglobin <9 g/dL
   6. Serum calcium >1.5 × ULN
   7. Total bilirubin > 2 × ULN
   8. Prothrombin time (PT) (International Normalized Ratio [INR]) >1.5 × ULN or activated partial thromboplastin time (aPTT) (sec) greater than the normal range
   9. Positive result for serum tests (hepatitis B or C virus, human immunodeficiency virus [HIV], rapid plasma reagin [RPR] test)
   10. Patients who show significant abnormalities in electrocardiogram (ECG) test results (e.g.,QTcF > 450 msec)
3. Subjects who received hypofractionated chemoradiation regimens (> 2 Gy per day)
4. Subjects with known hypersensitivity to components or excipients of clinical investigational drugs
5. Subjects with a history of drug abuse (especially hypnotics, centrally acting analgesics, opiates, or central nervous system drugs such as antipsychotic drugs)
6. Contraindicated Drugs and Treatments:

   1. Subjects who have administered cytochrome P450 (CYP) 3A4 or CYP2D6 inducers or inhibitors (e.g., carbamazepine, rifampin, ketoconazole, quinidine, fluoxetine, paroxetine, itraconazole, clarithromycin, etc.) within 28 days of baseline
   2. Subjects who received chemotherapy within 28 days of baseline (drugs or treatment known to have anticancer effects such as cytotoxic chemotherapy, antihormonal therapy, and targeted therapy)
   3. Subjects who have administered intravenous antibiotics, antivirals, or antifungals within 14 days from baseline
   4. Subjects who have administered benzodiazepines (e.g., lorazepam) within 3 days from baseline
   5. Subjects who participated in another clinical trial within 4 weeks of the baseline and administered the clinical trial drug
7. Subjects and their spouses (or partners) with childbearing potential who are not using medically acceptable methods of contraception for the duration of the trial and for 14 months (in female subjects) and 11 months (in male subjects) after the last dose of cisplatin treatment
8. Subjects who, in the judgment of other investigators, are not suitable to participate in the study"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) | 6 months and 12 months
  proportion of subjects who have a complete response (CR), partial response (PR), or stable disease (SD) at 6 months and 12 months will be summarized with the 95% confidence interval on the mITT and PP samples.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 6 months and 12 months
  The proportion of participants who achieve an ORR at 6 months and 12 months will be summarized with the 95% confidence interval on the mITT and PP samples.
Best overall response (BOR) | 6 months and 12 months
  The BOR will be based on all post-baseline disease assessments that occur prior to the initiation of subsequent anticancer therapy. BOR will be summarized for the following categories: CR, PR, SD, PD and non-evaluable.
Progression-free survival (PFS) | At 6 month and 1 year
  The PFS will be analyzed using Kaplan-Meier methods on the mITT and PP samples. KM estimates and associated two-sided 95% confidence intervals will be presented for each cohort. Participants who have no documented progression and are still alive at the time of analysis will be censored at the time of the latest date of assessment.
Locoregional control (LRC) | At 6 month and 1 year
  Rate of Locoregional recurrence after end of treatment (FDG-PET/CT scan).
Distant metastasis (DM) | through study completion, at most 1 year
  The proportion of participants who develop DM will be summarized with the 95% confidence interval on the mITT and PP samples
Overall survival (OS) | 1 year
  The OS will be analyzed using Kaplan-Meier methods on the mITT and PP samples. KM estimates and associated two-sided 95% confidence intervals will be presented for each cohort, and 1-year survival estimate will be calculated
Changes in tumor size | through study completion, at most 1 year
  Tumor imaging (CT and MRI) will be performed.
Number and severity of treatment-emergent adverse events (TEAEs), treatment-related AEs, and serious adverse events (SAEs) for all dose groups according to the NCICTCAE version 5.0 | through study completion, at most of 1 year
  AE will be measured by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Health-related quality of life (HR-QoL) | at week1, week8, week11, week 19, week 27 and week 52
  FACT-H&N V4.
  * Physical Well-Being
  * Social/Familiy Well-Being
  * Emotional Well-Being
  * Functinal Well-Being